CLINICAL TRIAL: NCT07383116
Title: A Randomized, Double-Blind, Multicenter Phase III Clinical Study of HB0025 Injection Combined With Chemotherapy Versus Tislelizumab Combined With Chemotherapy as First-Line Treatment for Locally Advanced or Metastatic Nonsquamous Non-Small Cell Lung Cancer
Brief Title: Phase III Clinical Study of HB0025 Combined With Chemotherapy Versus Tislelizumab Combined With Chemotherapy as First-Line Treatment for Advanced Nonsquamous Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Huaota Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HB0025-C-0303
Record Dates: First submitted 2026-01-15; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Non Squamous Non-small Cell Lung Cancer
Keywords: HB0025; Fist Line treatment; nonsq NSCLC
MeSH Terms: interventions — Pemetrexed; Carboplatin; Cisplatin; tislelizumab

STUDY DESIGN:
Intervention Model Description: This study plans to enroll approximately 500 subjects, who will be randomly assigned at a 1:1 ratio to either the HB0025 plus chemotherapy group (experimental group, ~250 subjects) or the tislelizumab plus chemotherapy group (control group, ~250 subjects). Subjects in the experimental group will receive HB0025 combined with chemotherapy, while those in the control group will receive tislelizumab combined with chemotherapy, with both regimens administered once every 3 weeks (Q3W). After completing 4 cycles of treatment, all subjects will proceed to the maintenance therapy phase with either HB0025 or tislelizumab plus pemetrexed (Q3W).
  Experimental group: HB0025 combined with pemetrexed plus carboplatin/cisplatin Control group: Tislelizumab combined with pemetrexed plus carboplatin/cisplatin
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HB0025 (Experimental): HB0025 combined with Pemetrexed for Injection plus Carboplatin for Injection or Cisplatin for Injection, intravenous infusion, once every 3 weeks (Q3W)
  Interventions: Drug: Pemetrexed injection; Drug: Carboplatin Injection; Drug: Cisplatin injection; Drug: HB0025 Injection
- Tislelizumab (Active Comparator): Tislelizumab combined with Pemetrexed for Injection plus Carboplatin for Injection or Cisplatin for Injection, intravenous infusion, once every 3 weeks (Q3W)
  Interventions: Drug: Pemetrexed injection; Drug: Carboplatin Injection; Drug: Cisplatin injection; Drug: Tislelizumab

INTERVENTIONS:
Drug: Pemetrexed injection — 500 mg/m², Q3W.
Drug: Carboplatin Injection — AUC 5, Q3W.
Drug: Cisplatin injection — 75 mg/m², Q3W.
Drug: HB0025 Injection — HB0025 Injection, ivgtt, Q3W，developed by Sponsor Huaota.
  Arms: HB0025
Drug: Tislelizumab — Tislelizumab, Active Control, intravenous infusion, once every 3 weeks (Q3W)
  Arms: Tislelizumab

SUMMARY:
This study is a randomized, controlled, double-blind, multicenter Phase III registration clinical trial, aiming to evaluate the efficacy and safety of HB0025 combined with chemotherapy (pemetrexed plus carboplatin/cisplatin) versus tislelizumab combined with chemotherapy (pemetrexed plus carboplatin/cisplatin) as a first-line treatment for unresectable locally advanced (Stage IIIB/IIIC) or metastatic (Stage IV) nonsquamous non-small cell lung cancer (NSCLC).

The study will take progression-free survival (PFS) assessed by Blinded Independent Central Review (BICR) as the primary endpoint, and plans to enroll approximately 500 subjects. After being eligible for screening, patients will be randomly assigned to the study groups at a ratio of 1:1 to receive either HB0025 combined with chemotherapy (experimental group) or tislelizumab combined with chemotherapy (control group). Both regimens will be administered once every 3 weeks (Q3W). After completing 4 cycles of treatment, patients will enter the maintenance therapy phase with HB0025 or tislelizumab plus pemetrexed (Q3W). The treatment will last until the investigator determines that there is no longer clinical benefit (based on comprehensive assessment of RECIST v1.1 imaging results and clinical symptoms), intolerable toxicity occurs, 35 cycles of study treatment are completed, or other treatment termination criteria specified in the protocol are met, whichever comes first.

DETAILED DESCRIPTION:
The random stratification factors of this study are as follows:

Disease stage (Stage IIIB/IIIC vs Stage IV); PD-L1 expression score indicator (Tumor Proportion Score, TPS): <1%, 1%-49%, ≥50%; Hepatic or brain metastasis (Yes vs No). This trial adopts the RECIST v1.1 criteria to conduct regular tumor response assessments for the subjects. Within 1 year (365 days) after the first dose, tumor assessments will be performed at Week 6 (±7 days), Week 12 (±7 days), and then every 9 weeks (±7 days) thereafter; after 1 year, assessments will be conducted every 12 weeks (±7 days).

If a subject discontinues study treatment due to reasons other than disease progression or death, tumor assessments should continue according to the fixed schedule until disease progression or study termination (whichever occurs later), initiation of new anti-tumor therapy, loss to follow-up, death, withdrawal of informed consent, or study completion, whichever occurs first.

At least 4 weeks after the first documentation of objective response, the objective response should be confirmed by re-assessment (in cases of clinical stability, the confirmation can be performed at the next scheduled assessment time point).

After the first documented radiological progression, if the investigator determines that the subject can still benefit from continued treatment and meets the criteria for continued treatment specified in the protocol, the subject may maintain the original treatment regimen until no clinical benefit is observed (assessed by the investigator).

If a subject withdraws from the study treatment due to reasons other than those mentioned above (e.g., occurrence of intolerable adverse events, completion of 24 months of HB0025 or tislelizumab treatment, or other reasons necessitating treatment discontinuation), a tumor assessment should be performed prior to study termination.

The investigator may conduct unscheduled tumor assessments (with an interval of at least 4 weeks from the previous assessment) when disease progression is suspected or other necessary circumstances arise. The sponsor will collect all imaging data of the subjects for BICR assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Able to fully understand and voluntarily sign the informed consent form, and willing and able to comply with the clinical study procedures and follow-up visits.
2. Aged 18 to 75 years old (inclusive of both upper and lower limits), male and female subjects are eligible.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-1.
4. Expected survival ≥ 12 weeks.
5. Histologically or cytologically confirmed locally advanced (Stage IIIB/IIIC) or metastatic (Stage IV) non-squamous non-small cell lung cancer (NSCLC) (confirmed per the 9th Edition of the TNM Staging System for Lung Cancer by the Union for International Cancer Control [UICC] and the American Joint Committee on Cancer [AJCC]), which is inoperable for radical resection and ineligible for radical concurrent/sequential chemoradiotherapy as well as immunotherapy as consolidation treatment.

   Note: For subjects with locally advanced (Stage IIIB/IIIC) non-squamous NSCLC who are inoperable for radical resection and ineligible for radical concurrent/sequential chemoradiotherapy as well as immunotherapy as consolidation treatment, assessment by relevant specialist physicians and provision of written documentation are required for confirmation.
6. No prior systemic antineoplastic treatment for the study disease (including systemic chemotherapy, targeted therapy, and immunotherapy).

   Note: Subjects who previously received neoadjuvant, adjuvant, or radical concurrent/sequential chemoradiotherapy for non-metastatic disease with curative intent are eligible if disease progression occurs > 180 days after the last dose of prior treatment.
7. Subjects must provide tumor tissue samples (archived or freshly obtained) collected at or after the diagnosis of locally advanced or metastatic tumor for central laboratory testing of PD-L1 expression.

   Note: The following samples are not accepted: fine-needle aspiration samples (without intact tissue structure, only cell suspensions or smears), brush cytology samples, cell smears from centrifuged pleural effusion drainage, bronchoalveolar lavage fluid samples, and bone lesions without soft tissue components or decalcified bone tumor samples. Tumor lesions used for fresh tissue biopsy should not be designated as RECIST v1.1 target lesions, unless the lesion is the only measurable lesion. For archived samples, they must be collected after the last systemic treatment, and the collection site must not have received radiotherapy. If a subject's archived samples do not meet the above requirements and the investigator judges that a biopsy is not in the subject's best interest, the use of archived samples may be permitted after discussion with the sponsor.
8. No sensitive EGFR mutations or ALK gene rearrangements. Prior tissue-based test reports for EGFR and ALK status must be provided. If the test reports do not meet the study requirements or are unavailable, tumor tissue samples must be provided for assessment of EGFR and ALK status (tested by a local laboratory recognized by the study site or the central laboratory) before enrollment.

   Note: For subjects with squamous NSCLC (excluding mixed-type NSCLC, e.g., adenosquamous carcinoma) who have a smoking history or are current smokers, if the prior EGFR and ALK status is unknown, testing for these markers is not required before enrollment, and they will be deemed negative.
9. Per RECIST v1.1 criteria (see Appendix 2), the subject must have at least one measurable (non-brain metastatic) lesion suitable for repeated and accurate measurement. Tumor lesions previously treated with radiotherapy or other local therapies must not be designated as target lesions, unless:

   The lesion is the only measurable lesion, and the investigator can provide imaging evidence (both pre- and post-local treatment) confirming clear disease progression of the lesion following local therapy; The lesion used for fresh tissue biopsy must not be designated as a target lesion, unless it is the only measurable lesion and the biopsy date is more than 4 weeks prior to the first dose of study treatment.
10. Confirmed adequate organ function, with mandatory compliance with the following laboratory parameters:

Hematology (no receipt of any blood component transfusion or hematopoietic growth factor support therapy within 14 days prior to screening tests):

1. Absolute Neutrophil Count (ANC) ≥ 1.5 × 10⁹/L;
2. Platelet Count (PLT) ≥ 100 × 10⁹/L;
3. Hemoglobin (HGB) ≥ 90 g/L;

Renal function:

1. Serum Creatinine (Scr) ≤ 1.5 × Upper Limit of Normal (ULN), and Creatinine Clearance (Ccr) ≥ 50 mL/min (calculated using the Cockcroft-Gault formula; see Appendix 3 for details);
2. Urine protein < 2+; if urine protein ≥ 2+, 24-hour urine protein excretion must be < 1 g;

Hepatic function:

1. Serum Total Bilirubin (TBiL) ≤ 1.5 × ULN; for subjects with liver metastasis or confirmed Gilbert's syndrome, TBiL ≤ 3 × ULN;
2. Serum Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 × ULN; for subjects with liver metastasis, ALT and AST ≤ 5 × ULN;
3. Serum Albumin (ALB) ≥ 30 g/L; Coagulation function: Activated Partial Thromboplastin Time (APTT) and International Normalized Ratio (INR) ≤ 1.5 × ULN (for subjects receiving anticoagulant therapy, the investigator must confirm that both INR and APTT are within the safe and effective therapeutic range); Cardiac function: Left Ventricular Ejection Fraction (LVEF) ≥ 50%. 11. Female and male subjects of childbearing potential must agree to use effective contraceptive measures from the screening period until 90 days after the last dose of study treatment. Discussion with the investigator is required to determine whether contraception can be discontinued after this period. Female subjects must not be breastfeeding. Female subjects of childbearing potential must have a negative serum pregnancy test result within 7 days before randomization.

Exclusion Criteria:

1. Histologically confirmed presence of any small cell carcinoma, neuroendocrine carcinoma, or sarcoma components [mixed-type NSCLC (e.g., adenosquamous carcinoma) is permitted for enrollment].
2. Known presence of driver gene alterations with approved first-line therapeutic options, such as sensitive EGFR mutations, ALK fusion, ROS1 fusion, BRAF V600 mutation, NTRK fusion, MET exon 14 skipping mutation, or RET fusion.
3. History of a second primary malignancy within 5 years before screening (enrollment is permitted for other malignancies cured by local treatment, e.g., carcinoma in situ of the cervix, localized cutaneous squamous cell carcinoma, basal cell carcinoma, ductal carcinoma in situ of the breast, < T1 urothelial carcinoma, and papillary microcarcinoma of the thyroid).
4. Symptomatic central nervous system (CNS) metastasis. For subjects with asymptomatic CNS metastasis or those with symptomatically stable CNS metastasis for ≥ 4 weeks prior to randomization, enrollment is permitted only if all the following criteria are met:

   * No metastasis to the meninges, midbrain, pons, medulla oblongata, spinal cord, or spinal cord compression; ② No increase in lesion size or new lesions after treatment;

     * No history of intracranial hemorrhage;

       * Discontinuation of corticosteroid therapy for ≥ 2 weeks prior to randomization; ⑤ No significant perilesional edema surrounding brain metastases; ⑥ The longest diameter of brain metastases ≤ 1.5 cm.
5. Prior receipt of immunotherapy, including immune checkpoint inhibitors (e.g., anti-PD-1/L1/L2, anti-CTLA-4 agents), immune checkpoint agonists (e.g., ICOS, CD40, GITR, OX40, CD137 agents), or cellular immunotherapy, or any treatment targeting the tumor immune mechanism. Additionally, for subjects who previously received PD-(L)1 inhibitors in the neoadjuvant/adjuvant setting or as consolidation therapy after definitive chemoradiotherapy, enrollment may be permitted (with sponsor approval) if the interval between the end of the last treatment and the occurrence of disease progression is more than 12 months.

   Note: For subjects with prior PD-(L)1 inhibitor exposure:

   Enrollment is prohibited if the subject experienced ≥ Grade 3 immune-related adverse events (irAEs) caused by prior immunotherapy (excluding endocrine-related irAEs), irAEs leading to permanent treatment discontinuation, ≥ Grade 2 immune-related cardiotoxicity, or immune-related neurological or ophthalmic irAEs of any grade; Screening is prohibited if all adverse events caused by prior immunotherapy have not been fully resolved or resolved to Grade 1 before study screening. For subjects with ≥ Grade 2 endocrine-related irAEs, enrollment is permitted if the condition is stable and asymptomatic with appropriate replacement therapy.
6. Prior receipt of systemic anti-angiogenic therapy, including but not limited to bevacizumab and its biosimilars, Endostar, small-molecule TKIs, and ramucirumab.
7. Prior anti-tumor therapy or concomitant medication (the washout period is calculated from the end date of the last treatment):a) Participation in any clinical trial within 28 days prior to the first dose;b) Receipt of anti-tumor therapy within 4 weeks prior to the first dose or within 5 half-lives of the drug (whichever is longer), including but not limited to chemotherapy, radiotherapy (thoracic radiotherapy with a dose > 30 Gy within 180 days prior to the first dose; non-thoracic radiotherapy with a dose > 30 Gy within 4 weeks prior to the first dose; local palliative radiotherapy with a dose ≤ 30 Gy for non-target lesions within 2 weeks prior to the first dose), targeted therapy, immunotherapy, or endocrine therapy;c) Use of Chinese herbal medicines (including patent Chinese medicines) with anti-tumor indications within 2 weeks prior to the first dose; use of non-specific immunomodulatory therapy (e.g., interleukin, interferon, thymosin, tumor necrosis factor, etc., excluding IL-11 for the treatment of thrombocytopenia) within 2 weeks prior to the first dose;d) Need for systemic administration of corticosteroids at a dose > 10 mg/day of prednisone or equivalent dose, or other immunomodulators within 2 weeks prior to randomization. [Short-term administration (≤ 7 days) for prophylaxis (e.g., contrast agent allergy) or treatment of non-autoimmune diseases (e.g., delayed hypersensitivity reaction caused by allergen exposure), or local administration (e.g., intraocular, intra-articular, intranasal, or inhaled administration) is permitted for enrollment];e) Use or current use of anticoagulants such as warfarin, heparin (excluding heparin for catheter locking or deep vein catheterization), dabigatran etexilate, rivaroxaban, etc., or antiplatelet drugs such as aspirin, clopidogrel, dipyridamole, cilostazol, or other known antiplatelet agents within 2 weeks prior to the first dose.
8. Major surgery or severe trauma within 4 weeks before the first dose of study treatment; inadequate recovery from prior surgery (as judged by the investigator); anticipated need for major surgery during the study; minor local surgery (e.g., needle biopsy, endoscopy, interventional procedure/examination, excluding vascular access establishment) within 7 days before randomization; presence of incompletely healed surgical incisions or wounds.
9. Active autoimmune disease requiring systemic treatment (e.g., treatment with immunomodulators or corticosteroids) within 2 years before screening, except for replacement therapy (e.g., thyroid hormone, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency).
10. Presence of any of the following infections:

    1. Severe infection (including but not limited to comorbidities requiring hospitalization, sepsis, or severe pneumonia) within 4 weeks before the first dose of study treatment; active infection requiring systemic anti-infective treatment (with antibiotics for ≥ 7 days) within 2 weeks before the first dose of study treatment;
    2. Known active tuberculosis (TB) (subjects with suspected active TB must undergo clinical examination to rule out the diagnosis);
    3. Known active syphilis infection;
    4. Has a known history of HIV;
    5. Active hepatitis B or hepatitis C; asymptomatic hepatitis B virus (HBV) carriers (HBV DNA ≤ 200 IU/ml or ≤ 1000 copies/ml or below the lower limit of detection, whichever is applicable) or subjects with clinically cured hepatitis C (HCV RNA below the lower limit of detection) are permitted for enrollment.

    Note: Anti-HBV treatment is required for HBsAg-positive subjects during the study treatment period.
11. Known hypersensitivity to protein drugs, recombinant proteins, components of HB0025, and/or components of chemotherapy drugs (pemetrexed and carboplatin/cisplatin).
12. Uncontrolled arterial hypertension despite standard treatment (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg).
13. Presence of any of the following severe comorbidities:

    1. Clinically significant bleeding (including but not limited to hemoptysis [defined as coughing up or expectorating ≥ 1 teaspoon (approximately 5 ml) of fresh blood or small blood clots, or hemoptysis without sputum; subjects with blood-tinged sputum or transient hemoptysis related to diagnostic bronchoscopy or lung biopsy are permitted], gastrointestinal bleeding, nasal bleeding [subjects with bloody nasal discharge are permitted]) within 4 weeks before the first dose of study treatment; any arterial thrombosis or embolism event, or significant vascular disease (e.g., aortic aneurysm, aortic dissection) within 180 days before the first dose of study treatment; history of deep vein thrombosis within 90 days before the first dose of study treatment;
    2. Imaging findings at screening showing: Tumor invasion of large blood vessels (e.g., central pulmonary artery, central pulmonary vein, aorta, brachiocephalic artery, common carotid artery, subclavian artery, superior vena cava); tumor invasion of vital organs (e.g., heart, trachea, esophagus, main bronchus); or imaging evidence of risk for esophagotracheal fistula or esophagopleural fistula; tumor encasement of large blood vessels with vascular stenosis; or pulmonary lesions with obvious necrosis/cavitation (as judged by the investigator to pose a bleeding risk if enrolled);
    3. History of persistent bleeding disorders or coagulation disorders (past or current);
    4. Clinically significant (e.g., active) cardiovascular or cerebrovascular disease within 180 days prior to the first dose, including but not limited to unstable angina requiring hospitalization, myocardial infarction, myocarditis, cardiomyopathy, congestive heart failure of New York Heart Association (NYHA) Class ≥ III, poorly controlled severe arrhythmia, transient ischemic attack (TIA), cerebrovascular accident (CVA), or vascular disease (e.g., aortic aneurysm at risk of rupture); or other cardiac impairment that may affect the safety evaluation of the study drug (e.g., poorly controlled arrhythmia, myocardial ischemia). Prolonged Fridericia-corrected QT interval (QTcF) on electrocardiogram: > 450 ms for males and > 470 ms for females.
    5. History of conditions potentially causing gastrointestinal bleeding or perforation (e.g., gastrointestinal obstruction, acute Crohn's disease, ulcerative colitis, esophagogastric varices, gastrointestinal perforation, unhealed wound, intra-abdominal abscess, or acute gastrointestinal bleeding) within 180 days before the first dose of study treatment; subjects with chronic Crohn's disease or ulcerative colitis (excluding those who have undergone total colectomy and proctectomy) are excluded, even if in remission;
    6. History of gastrointestinal fistula or genitourinary fistula (past or current) that remains unhealed after surgical treatment;
    7. Hydronephrosis unrelieved by nephrostomy or ureteral stenting, or infected hydronephrosis/hydroureter;
    8. Current presence of third-space fluid collections (e.g., pleural effusion, pericardial effusion, abdominal/pelvic effusion) requiring repeated puncture/drainage for local management; or receipt of local drainage within 2 weeks before the first dose of study treatment;
    9. Acute exacerbation of chronic obstructive pulmonary disease within 30 days before the first dose of study treatment;
    10. Current presence of uncontrolled comorbidities, including but not limited to decompensated liver cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, severe active peptic ulcer disease or gastritis (enrollment decision requires joint discussion between the investigator and the sponsor).
14. Current presence of interstitial lung disease, pneumoconiosis, or drug/radiotherapy-related pneumonia requiring treatment.
15. Unresolved adverse events from prior treatment (defined as adverse events not resolved to Grade 0 or 1 per the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 5.0, or to the level specified in the inclusion/exclusion criteria), except for alopecia. Subjects with irreversible toxicity (e.g., hearing loss) that is not expected to worsen after administration of study drugs may be enrolled after consultation with the medical monitor. Subjects with long-term radiotherapy-induced toxicity (judged by the investigator as irreversible) may be enrolled after consultation with the medical monitor.
16. Pregnancy, lactation, or plans to breastfeed during the study.
17. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
18. Receipt of live virus vaccines or attenuated live vaccines within 30 days before randomization, or planned vaccination during the study (Note: Inactivated vaccines are permitted).
19. Known history of mental illness, alcoholism, drug addiction, or substance abuse.
20. Past or current presence of uncontrolled metabolic disorders, non-tumor-related local/systemic diseases, tumor-induced diseases or symptoms (e.g., cachectic manifestations: weight loss > 10% within 3 months before screening), laboratory abnormalities, or any treatment that may pose a high medical risk, confound study results, interfere with the subject's full participation in the study, or make study participation not in the subject's best interest.
21. Subjects deemed unsuitable for study participation by the investigator for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-04-10 (Estimated); Study Completion 2028-04-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 Months
  PFS is defined as the time from the date of randomization till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first)

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 24 Months
  OS is defined as the period from the start of randomization to the time of death due to any cause according to RECIST 1.1.
Objective Response Rate (ORR) | Up to 24 Months
  ORR is defined as the proportion of subjects achieving the best overall therapeutic effect (BOR) as complete remission (CR) or partial remission (PR) according to RECIST 1.1 by investigator.
Disease control rate (DCR) | Up to 24 Months
  DCR defined as the number of patients were confirmed CR and/or PR and/or stable disease(SD) according to RECIST 1.1 by investigator divided by the patients with at least one tumour evaluation
Duration of response (DOR) | Up to 24 Months
  DOR is defined as the time from the first record of CR or PR to the first record of disease. DOR as evaluated by investigators according to RECIST v1.1.
Time to Progression(TTP) | Up to 24 Months
  TTP is defined as the time from the time of randomization to the occurrence of disease progression according to recist 1.1 by investigator.
Objective Response Rate (ORR)-BICR | Up to 24 Months
  ORR is defined as the proportion of subjects achieving the best overall therapeutic effect (BOR) as complete remission (CR) or partial remission (PR) according to RECIST 1.1 by BICR
Disease control rate (DCR)-BICR | Up to 24 Months
  DCR defined as the number of patients were confirmed CR and/or PR and/or stable disease(SD) according to RECIST 1.1 by BICR divided by the patients with at least one tumour evaluation
Duration of response (DOR)-BICR | Up to 24 Months
  DOR is defined as the time from the first record of CR or PR to the first record of disease. DOR as evaluated by BICR according to RECIST v1.1
Time to Progression(TTP)-BICR | Up to 24 Months
  TTP is defined as the time from the time of randomization to the occurrence of disease progression according to recist 1.1 by BICR
Safety Assement | Up to 24 Months
  The incidence, severity and outcome of adverse events (AE), serious adverse events (SAE), immune-related adverse events (irAE) and adverse events of special concern (AESI) per NCI-CTCAE V5.0
Maximum serum concentration(Cmax) | Up to 24 Months
  Cmax refers to The maximum blood concentration of HB0025 after administration. - Sample concentration analysis method adopts ELISA. parameters will be calculated by Phoenix WinNonlin version 8.3.
Anti-drug antibodies (ADA) | Up to 24 Moths
  Incidence of positive anti-drug antibodies(ADA).

OTHER OUTCOMES:
PD-L1 expression | Approximately 16 months.
  Exploring the correlation between the levels of biomarkers (PD-L1) and the efficacy of combined treatment by Immunohistochemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, MD, Principal Investigator — The East Hospital Affiliated to Tongji University, Shanghai, Shanghai 200120
Locations (1):
- The East Hospital Affiliated to Tongji University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided